CLINICAL TRIAL: NCT06382753
Title: Impact of Periodontal Supportive Therapy Number of Sessions in Patients With Gingivitis and Periodontitis in Order to Evaluate Disease Evolution.
Brief Title: Impact of Periodontal Supportive Therapy in Patients With Gingivitis and Periodontitis
Status: Recruiting | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Associate Professor, University of Catania
Other Study IDs: 20-24-PAR
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Gingivitis; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gingival inflammation — Patients were scored for their status of gingival inflammation using Gingival Index and Bleeding on Probing Scores

SUMMARY:
The study evaluated the number of sessions of periodontal supportive treatment in patients with gingivitis in order to evaluate the risk of periodontitis development.

DETAILED DESCRIPTION:
Patient with gingivitis were retrospectively evaluated. The number of periodontal supportive therapy were recorded other than gingivitis periodontal parameters over 5-years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gingivitis

Exclusion Criteria:

* Diagnosis of Periodontitis
* Pregnancy
* Systemic diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 patients with diagnosed gingivitis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding on Probing | 5-years
  Evaluation of bleeding on probing reduction

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 1-year
Access Criteria: Pubmed
URL: http://pubmed.gov